CLINICAL TRIAL: NCT06832852
Title: Is a Stepped Model of Care Cost-effective Compared to Usual Care for Musculoskeletal Disorders? a Randomized Controlled Trial
Brief Title: Which Model of Care is the Most Cost-effective in the Treatment of Musculoskeletal Disorders?
Acronym: Edu1st
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 495615
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Neck Pain; Anterior Knee Pain Syndrome; Rotator-cuff Related Shoulder Pain
Keywords: Stepped-Care; Rehabilitation; Musculoskeletal Disorders; Education; Medical Care
MeSH Terms: conditions — Low Back Pain; Neck Pain; Patellofemoral Pain Syndrome; Musculoskeletal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given that for the type of intervention provided, it is impossible to blind the care provider and participants, only the statistician and outcome assessors will be blinded. All groups will be treated in different clinics to reduce potential contamination: Usual Medical Care in FP Clinics and the Stepped Care and the Usual Rehabilitation Care in different PT clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stepped Care Group (Experimental): During the first 6 weeks, participants will take part in a self-management education program and will be offered two individual educational sessions provided by a physiotherapist (PT). At the 6-week follow-up evaluation, the score on a region-specific patient-reported outcome measure will be used to determine if the condition is resolved or unresolved. Those no longer experiencing clinically important symptoms at the 6-week follow-up will be considered resolved and will have no further intervention. Those with remaining clinically important symptoms will receive follow-up interventions by a PT with up to 5 sessions over 6 weeks. The rehabilitation program will be similar to the one received by the participants in the Usual Rehabilitation Care Group.
  Interventions: Other: Stepped care
- Usual Rehabilitation Care Group (Active Comparator): Participants will take part in a pragmatic 12-week physiotherapist (PT)-led rehabilitation program. It will include a maximum of 10 supervised meetings of 30 minutes each and an individualized home exercise program of 20-30 minutes to be performed 3-4 times per week.
  Interventions: Other: Rehabilitation Care
- Usual Medical Care Group (Active Comparator): Participants will take part in a 12-week family physician (FP)-led program based on best practices and CPGs. It will include a maximum of 3 meetings over 12 weeks with a FP.
  Interventions: Other: Medical Care

INTERVENTIONS:
Other: Stepped care — During the first education session, participants will be provided with information pertaining to painful area, basic pain science, injury specific advice on load management, pain and activity management, lifestyle factors and physical activity. A general physical activity will be recommended (150-300 minutes of moderate-intensity activity per week). Then, participants will be directed to a website developed by the research team and patient partners. The website includes explanations of the various topics discussed during the session , explanatory videos, and summarized information. During the second educational session, the participant's condition will be reviewed, and their understanding of the topics covered in the first session and on the website will be assessed. A follow-up on the website will also be conducted. The physiotherapist will then answer the participant's questions and provide personalized advice based on their condition, along with long-term recommendations.
  Arms: Stepped Care Group
Other: Rehabilitation Care — The pragmatic rehabilitation program will include exercises aimed at improving strength, endurance, flexibility, capacity to sustain mechanical load and dynamic control. Manual therapy may be provided during the sessions, based on pragmatic clinical decision-making. Participants will also receive information pertaining to the painful area and advice on pain and load management, and on activity modification, integrated across the sessions.
  Arms: Usual Rehabilitation Care Group
Other: Medical Care — The pragmatic medical intervention may include pharmacological management, education, physiotherapy referral or referral to a specialist as deemed necessary.
  Arms: Usual Medical Care Group

SUMMARY:
As musculoskeletal disorders (MSKDs) reach epidemic proportions in Canada, access to the public health system for those who suffer from them is increasingly difficult. One of the main barriers is the delays to see a publicly funded health professional. New models of care must therefore be developed to ensure better access. We have previously shown that not all patients with a MSKD need to be closely followed by a health professional as for a large proportion of patients simply educating them is enough to resolve their MSKD. A stepped care model where education would be given first before deciding if patients need a more extensive follow-up should be explored. This project will compare the effectiveness of a Stepped Care Model to that of the two most widely used models of care: Usual Medical Care and Usual Rehabilitation Care. We think that a Stepped Care Model will be as effective to reduce functional limitations, but will lead to lower healthcare costs.

Adults (n=369) with a MSKD will be randomly assigned to one of the intervention groups: Stepped Care, Usual Medical Care (physician-led intervention: e.g., advice/education, pharmacological pain management), or Usual Rehabilitation Care (physiotherapist-led intervention: e.g., advice/education, exercises). Participants in the Stepped Care Group will take part in two education sessions during the first 6 weeks. After 6 weeks, those who still have clinically important symptoms will receive follow-up rehabilitation interventions, while those who don't will be considered recovered and will have no further intervention. Primary (functional limitations) and secondary (e.g., pain, quality of life) outcomes will be assessed at baseline, and at 6, 12 and 24 weeks, and costs estimate will be established for each model of care. Knowing the urgent need for an overhaul of services to reduce wait times, the Stepped Care Model proposed could be a solution to improve access to health services without compromising quality of care.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSKDs) are a leading cause of global disability, pain and work disability. Even if they are not fatal, they are disabling and their care places a significant burden on the healthcare system. Knowing that early intervention improves clinical outcomes, the healthcare system must ensure that those affected have access to the care they need, which is currently not the case. Optimizing the use of resources through the development of innovative and effective interventions must therefore be addressed. In randomized controlled trials (RCTs) conducted by our team, we have demonstrated that not all patients with MSKDs need to be closely followed by a health professional as for a large proportion of patients simply educating them is enough to resolve their MSKD. As healthcare costs escalate, using a Stepped Care Model in which patient education is offered first, providing usual care only to those whose symptoms have not resolved might lead to more efficient healthcare use and lower costs. The primary objective of this RCT is to establish the effectiveness of a new model of care for MSKDs by comparing a Stepped Care Model to the two most widely used models of care: Usual Medical Care and Usual Rehabilitation Care. A secondary objective will be to compare the costs associated with each of these care models. We hypothesize that a Stepped Care Model will be as effective as Usual Medical and Rehabilitation Care to reduce functional limitations, but will lead to lower costs.

In this pragmatic parallel-group RCT, 369 adults presenting a MSKDs will be randomly assigned to one of the intervention groups: 1) Stepped Care, 2) Usual Medical Care (physician-led intervention [up to 3 appointments within 12 weeks]: e.g., advice/education, pharmacological pain management), 3) Usual Rehabilitation Care (physiotherapist-led intervention [up to 10 appointments within 12 weeks]: e.g., advice/education, exercises). During the first 6 weeks of the study, participants in the Stepped Care Group will take part in a self-management education program that includes two education sessions with a physiotherapist; after 6 weeks, those still experiencing clinically important symptoms will receive follow-up rehabilitation interventions (up to 5 sessions within 6 weeks), while those not experiencing clinically important symptoms will be considered recovered and will have no further intervention. The primary (functional limitations) and secondary outcomes (e.g., pain severity, health-related quality of life, pain-related fear, pain self-efficacy), assessed at baseline and at 6, 12 and 24 weeks, will be compared between the groups using repeated measures analyses (linear mixed models). Costs estimate from the public payer and patient perspective will be established (including incremental cost-effectiveness and cost-utility ratios) and compare between care models (one-way ANOVA). Our research team has all the expertise (health services organization, medicine, rehabilitation, biostatistics, health economics) necessary to carry out this project. Knowing the urgent need for an overhaul of services to reduce wait times and ensure equitable access, the Stepped Care Model proposed could be a solution to improve access to health services without compromising quality of care. If the results are conclusive, they would lay the foundation for a future pan-Canadian trial examining the benefits of implementing such a model into the public healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* present with one of the four targeted MSKDs (low back pain, neck pain, anterior knee pain, rotator cuff-related shoulder pain).
* have had pain for at least 6 weeks.
* For low back pain (LBP): 1) non-specific LBP with or without radiation to the lower limbs, 2) minimal score of 15 on the ODI.
* For neck pain : 1) non-specific neck pain with or without radiation to the upper limbs, 2) minimal score of 21 on the NDI.
* For anterior knee pain : 1) anterior knee pain during walking, running or going up or down stairs, or during at least two activities among: kneeling, squatting, and resisted knee extension, 2) maximum score of 79 on the KOS-ADL.
* For rotator cuff-related shoulder pain : 1) minimal score of 15 on the QuickDASH, and 2) shoulder pain attributed to a rotator cuff-related shoulder pain using diagnostic guidelines of the British Elbow and Shoulder Society.

Exclusion Criteria:

* Unavailable to participate during the 24 weeks of the study.
* Do not understand French or English.
* Diagnosis of rheumatoid, inflammatory or neurodegenerative diseases.
* Received a corticosteroid injection in the previous 3 months.
* Cognitive problems interfering (Mini-Mental State Examination ≥ 24).
* Received a corticosteroid injection in the previous 3 months.
* Less than 6 weeks since an intervention for their condition (including performing prescribed condition-specific exercises or taking prescribed medication).
* For low back pain (LBP): 1) LBP related to specific conditions (e.g., vertebral fracture, infections, neuropathic pain [>4 at the DN4 questionnaire]), 2) history of spine surgery or signs of upper motor neuron lesions (bilateral paresthesia, hyperreflexia or spasticity)..
* For neck pain : 1) neck pain related to specific conditions (e.g.; vertebral fracture, infections, neuropathic pain [>4 at the DN4 questionnaire]), 2) history of spine surgery or signs of upper motor neuron lesions.
* For anterior knee pain : 1) history of knee surgery or patellar dislocation, 2) pain believed to originate either from meniscus or from any knee ligament.
* For rotator cuff-related shoulder pain : 1) history of shoulder surgery, dislocations, fractures or capsulitis, 2) full thickness rotator cuff tear identified by imagery or clinical tests (lag signs and gross weakness).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional limitations | 24 weeks after baseline
  Functional limitations will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain.

SECONDARY OUTCOMES:
Functional limitations | 6 weeks after baseline
  Functional limitations will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain.
Functional limitations | 12 weeks after baseline
  Functional limitations will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain.
Pain Severity | 6 weeks after baseline
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity.
Pain Severity | 12 weeks after baseline
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity.
Pain Severity | 24 weeks after baseline
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity.
Health-related quality of life | 6 weeks after baseline
  Health-related quality of life will be measured using the EQ-5D-5L. EQ-5D-5L is a 5-item generic HRQoL questionnaire covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score.
Health-related quality of life | 12 weeks after baseline
  Health-related quality of life will be measured using the EQ-5D-5L. EQ-5D-5L is a 5-item generic HRQoL questionnaire covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score.
Health-related quality of life | 24 weeks after baseline
  Health-related quality of life will be measured using the EQ-5D-5L. EQ-5D-5L is a 5-item generic HRQoL questionnaire covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score.
Pain-related fear | 6 weeks after baseline
  Pain-related fear will be evaluated using the Tampa Scale for Kinesiophobia. The Tampa Scale for Kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging.
Pain-related fear | 12 weeks after baseline
  Pain-related fear will be evaluated using the Tampa Scale for Kinesiophobia. The Tampa Scale for Kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging.
Pain-related fear | 24 weeks after baseline
  Pain-related fear will be evaluated using the Tampa Scale for Kinesiophobia. The Tampa Scale for Kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging.
Pain catastrophizing | 6 weeks after baseline
  Pain catastrophizing will be evaluated using the Pain Catastrophizing Scale. The Pain Catastrophizing Scale is a 13-item scale aiming to identify catastrophic thoughts about pain.
Pain catastrophizing | 12 weeks after baseline
  Pain catastrophizing will be evaluated using the Pain Catastrophizing Scale. The Pain Catastrophizing Scale is a 13-item scale aiming to identify catastrophic thoughts about pain.
Pain catastrophizing | 24 weeks after baseline
  Pain catastrophizing will be evaluated using the Pain Catastrophizing Scale. The Pain Catastrophizing Scale is a 13-item scale aiming to identify catastrophic thoughts about pain.
Pain self-efficacy | 6 weeks after baseline
  Pain self-efficacy will be evaluated using the Pain Self-Efficacy Questionnaire. The Pain Self-Efficacy Questionnaire consists of 10 items utilized to measure patient's confidence in performing daily activities despite of pain.
Pain self-efficacy | 12 weeks after baseline
  Pain self-efficacy will be evaluated using the Pain Self-Efficacy Questionnaire. The Pain Self-Efficacy Questionnaire consists of 10 items utilized to measure patient's confidence in performing daily activities despite of pain.
Pain self-efficacy | 24 weeks after baseline
  Pain self-efficacy will be evaluated using the Pain Self-Efficacy Questionnaire. The Pain Self-Efficacy Questionnaire consists of 10 items utilized to measure patient's confidence in performing daily activities despite of pain.
Anxiety and depressive symptoms | 6 weeks after baseline
  Anxiety and depressive symptoms will be measured using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale is a 14-item self-administered questionnaire used to screen the presence of depression and anxiety.
Anxiety and depressive symptoms | 12 weeks after baseline
  Anxiety and depressive symptoms will be measured using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale is a 14-item self-administered questionnaire used to screen the presence of depression and anxiety.
Anxiety and depressive symptoms | 24 weeks after baseline
  Anxiety and depressive symptoms will be measured using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale is a 14-item self-administered questionnaire used to screen the presence of depression and anxiety.
Region-specific symptoms and functional limitations - Low back pain | 6 weeks after baseline
  The modified Oswestry Disability Index is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living. The modified Oswestry Disability Index will only be filled by participants with low back pain.
Region-specific symptoms and functional limitations - Low back pain | 12 weeks after baseline
  The modified Oswestry Disability Index is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living. The modified Oswestry Disability Index will only be filled by participants with low back pain.
Region-specific symptoms and functional limitations - Low back pain | 24 weeks after baseline
  The modified Oswestry Disability Index is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living. The modified Oswestry Disability Index will only be filled by participants with low back pain.
Region-specific symptoms and functional limitations - Neck pain | 6 weeks after baseline
  The Neck Disability Index is a 10-item questionnaire that measures a patient's self-reported neck pain-related disability. The Neck Disability Index will only be filled by participants with neck pain.
Region-specific symptoms and functional limitations - Neck pain | 12 weeks after baseline
  The Neck Disability Index is a 10-item questionnaire that measures a patient's self-reported neck pain-related disability. The Neck Disability Index will only be filled by participants with neck pain.
Region-specific symptoms and functional limitations - Neck pain | 24 weeks after baseline
  The Neck Disability Index is a 10-item questionnaire that measures a patient's self-reported neck pain-related disability. The Neck Disability Index will only be filled by participants with neck pain.
Region-specific symptoms and functional limitations - Rotator cuff-related shoulder pain | 6 weeks after baseline
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. The QuickDASH will only be filled by participants with rotator cuff-related shoulder pain.
Region-specific symptoms and functional limitations - Rotator cuff-related shoulder pain | 12 weeks after baseline
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. The QuickDASH will only be filled by participants with rotator cuff-related shoulder pain.
Region-specific symptoms and functional limitations - Rotator cuff-related shoulder pain | 24 weeks after baseline
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. The QuickDASH will only be filled by participants with rotator cuff-related shoulder pain.
Region-specific symptoms and functional limitations - Anterior knee pain | 6 weeks after baseline
  The Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS) is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations. The KOS-ADLS will only be filled by participants with anterior knee pain.
Region-specific symptoms and functional limitations - Anterior knee pain | 12 weeks after baseline
  The Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS) is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations. The KOS-ADLS will only be filled by participants with anterior knee pain.
Region-specific symptoms and functional limitations - Anterior knee pain | 24 weeks after baseline
  The Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS) is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations. The KOS-ADLS will only be filled by participants with anterior knee pain.
Health costs | 12 weeks after baseline
  Health costs will be estimated using the CoPaQ. The CoPaQ measures patients' costs, including those of informal caregivers. It includes questions on costs associated with treatments such as copays, transport to sessions, child care, time off work, and loss in revenue.
Health costs | 24 weeks after baseline
  Health costs will be estimated using the CoPaQ. The CoPaQ measures patients' costs, including those of informal caregivers. It includes questions on costs associated with treatments such as copays, transport to sessions, child care, time off work, and loss in revenue.
Healthcare resource utilization | 12 weeks after baseline
  Healthcare resource utilization will be estimated using a ressource utilization questionnaire. The questionnaire will include questions on appointment with family physicians, physiotherapists or any other health professionals, medical imaging, laboratory tests, pain medication and indirect.
Healthcare resource utilization | 24 weeks after baseline
  Healthcare resource utilization will be estimated using a ressource utilization questionnaire. The questionnaire will include questions on appointment with family physicians, physiotherapists or any other health professionals, medical imaging, laboratory tests, pain medication and indirect.
Participants' satisfaction with their condition | 6 weeks after baseline
  Participants' satisfaction with their condition will be assessed using the Patient Acceptable Symptom State (PASS). It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.96
Participants' satisfaction with their condition | 12 weeks after baseline
  Participants' satisfaction with their condition will be assessed using the Patient Acceptable Symptom State (PASS). It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.96
Participants' satisfaction with their condition | 24 weeks after baseline
  Participants' satisfaction with their condition will be assessed using the Patient Acceptable Symptom State (PASS). It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.96
Satisfaction with treatment received | 12 weeks after baseline
  Participants will rate their satisfaction with treatment received ("not satisfied'', "satisfied'', "very much satisfied''), with the duration of treatments ("too short'', "long enough'', "too long''), with the frequency of treatments and with the time spent with the health professional during treatments ("not enough'', "just right'', "too much'') using a 3-item Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- Centre for interdisciplinary research in rehabilitation and social integration (Cirris), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are awaiting confirmation from the ethics research committee regarding permission to share individual participant data with other researchers. Once confirmed, we will outline the plan.

REFERENCES:
- [Derived] Roy JS, Masse-Alarie H, Dube MO, Pinard AM, Lamontagne M, Sole G, Tittley J, Laberge M, Dupuis F, Fiset F, Nduwimana I, McArthur E, Desmeules F. Effectiveness and Cost-Effectiveness of a Stepped Model of Care for Musculoskeletal Disorders: Protocol for a Multiarm Randomized Controlled Trial (Edu-First Trial). JMIR Res Protoc. 2025 Nov 19;14:e77574. doi: 10.2196/77574. PMID 41258669